CLINICAL TRIAL: NCT06249048
Title: A Phase 1/2, Open-label, Multi-center, First-in-human Study of the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics and Anti-tumor Activity of STX-001 Delivered by Intratumoral Injection in Patients With Advanced Solid Tumors as a Monotherapy or in Combination With Pembrolizumab
Brief Title: Phase 1/2 Study of Intratumoral Injection of STX-001 in Advanced Solid Tumors as Monotherapy or in Combination With Pembrolizumab
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Strand Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STX-001-01
Record Dates: First submitted 2024-02-02; First posted 2024-02-08 (Actual); Last update posted 2025-10-29 (Actual); Status verified 2025-10

CONDITIONS: Advanced Solid Tumor
Keywords: Intratumoral; Triple Negative Breast Cancer; Melanoma; Advance Solid Tumors; mRNA
MeSH Terms: conditions — Triple Negative Breast Neoplasms; Melanoma | interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Phase 1 Monotherapy (STX-001) (Experimental): A Phase 1, first-in-human (FIH), multiple ascending dose administration of intratumoral STX-001 monotherapy to evaluate safety, tolerability, pharmacokinetics (PK), pharmacodynamics (PD) and preliminary antitumor activity in patients with advanced cancers. Consists of four planned dose-escalation cohorts (Cohorts 1m) plus permitted backfill enrollment (up to 30 patients). New patients are enrolled in each dose escalation cohort, and dose escalation may be stopped early if emerging PK or safety data warrant it. Dose extension and treatment pauses are integrated, with a maximum extension of 35 cycles (≈24 months).
  Interventions: Biological: STX-001
- Phase 1 Combination (STX-001 with Pembrolizumab) (Experimental): A Phase 1, first-in-human (FIH), multiple ascending STX-001 dose administration, in combination with pembrolizumab, to evaluate the safety, tolerability, pharmacokinetics (PK), pharmacodynamics (PD), and preliminary antitumor activity in patients with advanced cancers. Consists of 4 planned dose escalation cohorts (Cohorts 1c) of STX-001and pembrolizumab given concurrently, with new patients enrolled in each dose escalation cohort. Dose escalation may be halted early if PK or safety data indicate, and the dose extension period extends up to 35 cycles with treatment pauses. Backfill enrollment is permitted up to 30 patients.
  Interventions: Biological: STX-001; Biological: Keytruda®
- Phase 2 Combination (STX-001 with Pembrolizumab) (Experimental): Phase 2 consists of dose expansion cohorts in patients with 2 defined cancer types: triple negative breast cancer (TNBC) and melanoma. Phase 2 will evaluate STX-001 in combination with pembrolizumab; the recommended Phase 2 dose (RP2D) of STX-001 will be selected based on analysis of the totality of data from Phase 1 safety, tolerability, pharmacokinetics (PK), pharmacodynamics (PD) and preliminary efficacy data. Dose extension and treatment pauses are incorporated.
  Interventions: Biological: STX-001; Biological: Keytruda®
- Phase 1 Visceral-lesion Monotherapy (Cohort 1Vm) (Experimental): Phase 1, first-in-human (FIH) monotherapy cohort targeting visceral lesions. STX-001 is administered intratumorally at 30 µg, 100 µg and 300 µg to evaluate safety, tolerability, pharmacokinetics (PK), pharmacodynamics (PD), and preliminary antitumor activity in patients with advanced cancers. Cohort 1Vm is part of the dose escalation stage; new patients are enrolled at each dose level, and backfill enrollment is permitted up to 30 patients. Dose escalation may be stopped early if PK or safety data warrant it.
  Interventions: Biological: STX-001
- Phase 2 Advanced-Melanoma Monotherapy (Experimental): Phase 2 dose expansion cohort evaluating STX-001 monotherapy administered intratumorally to patients with advanced melanoma. Assesses safety, tolerability, pharmacokinetics (PK), pharmacodynamics (PD), and preliminary antitumor activity with the recommended dose selected based on Phase 1 data. Dose extension and treatment pauses are allowed up to 35 cycles.
  Interventions: Biological: STX-001

INTERVENTIONS:
Biological: STX-001 — STX-001 encapsulates a self-replicating RNA encoded for IL-12, contained within an LNP for intratumoral injection. Injections may be administered into multiple lesions according to protocol-defined procedures.
Biological: Keytruda® — Pembrolizumab (Keytruda USPI 2023) is a marketed PD-1 blocking humanized monoclonal IgG4 kappa antibody.
  Other Names: Pembrolizumab
  Arms: Phase 1 Combination (STX-001 with Pembrolizumab); Phase 2 Combination (STX-001 with Pembrolizumab)

SUMMARY:
Phase 1/2, Open-label, Multi-center, First-in-human Study of the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics and Anti-tumor Activity of STX-001 Delivered by Intratumoral Injection in Patients with Advanced Solid Tumors as a Monotherapy or in Combination with Pembrolizumab. The study now includes a monotherapy cohort targeting visceral lesions and a separate Phase 2 monotherapy cohort for advanced melanoma.

DETAILED DESCRIPTION:
This open-label, Phase 1/2, first-in-human (FIH), multiple ascending dose and dose expansion study involves STX-001 administration, alone or in combination with pembrolizumab, to evaluate the safety, tolerability, pharmacokinetics (PK), pharmacodynamics (PD), and preliminary antitumor activity in patients with advanced cancers.

Phase 1 consists of 4 planned dose escalation cohorts of STX-001 delivered as a monotherapy (Cohorts 1m), 4 planned dose escalation monotherapy cohorts of STX-001 delivered as a combination therapy with pembrolizumab treatment given concurrently (Cohorts 1c), and an additional monotherapy cohort targeting visceral lesions (Cohort 1vm) that will be evaluated at 30ug, 100ug and 300ug. New patients will be enrolled in each dose escalation cohort.

Phase 2 consists of dose expansion cohorts in patients with 2 defined cancer types: triple-negative breast cancer (TNBC) and melanoma. There will also be a monotherapy cohort for advanced melanoma. Phase 2 will evaluate STX-001 in combination with pembrolizumab; the recommended Phase 2 dose (RP2D) will be selected based on analysis of the totality of data from Phase 1 safety, tolerability, PK, PD and preliminary efficacy data.

ELIGIBILITY:
General Inclusion Criteria:

* ≥ 18 years of age at the time of screening.
* Mentally competent and able to understand and sign the informed consent form (ICF).
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
* Life expectancy of ≥ 12 weeks per the Investigator.
* Body weight ˃ 40 kg.
* At least 4 weeks from any prior major surgery.
* Willing and able to provide blood samples prior to the start of this study.
* Has a tumor lesion amenable to injection, must be accessible for pre and post injection biopsy, and the patient must be willing to consent to biopsy, if deemed safe by the Investigator.
* Laboratory values (Hematology): Absolute neutrophil count ≥ 1,000 cells/mm3; Platelet count ≥ 75,000 cells/mm3; Hemoglobin ≥ 8.0 g/dL.
* Laboratory values (Renal): Serum creatinine < 1.5 × upper limit of normal (ULN) or creatinine clearance ≥ 40 mL/min based on the Cockcroft-Gault glomerular filtration rate estimation
* Laboratory values (Coagulation): Prothrombin/International Normalized Ratio (PT/INR) or prothrombin time must be < 1.5 × ULN;
* Activated partial thromboplastin time (aPTT) ≤ 1.5 × ULN unless undergoing anticoagulation therapy.
* Laboratory values (Liver): Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) < 2 × ULN; Bilirubin ≤ 2 × ULN or ≤ 5 × ULN for all patients.

Phase 1 Inclusion Criteria:

* Histologically or cytologically documented, locally advanced, or metastatic solid tumor.
* Disease progression confirmed by imaging or other objective evidence after having received standard treatment or patients with refractory solid tumors. Patients must have progressed or are intolerant of at least one line of prior therapy.

Phase 2 Inclusion Criteria (TNBC):

* Histologically or cytologically documented findings consistent with TNBC not amenable to curative surgery, radiation, or other therapy.
* Prior treatment (for advanced, metastatic or [neo]adjuvant) should have included a taxane and/or anthracycline-based therapy and, where appropriate, an approved checkpoint inhibitor.
* Has disease other than the injected lesion that is measurable by RECIST 1.1.

Phase 2 Inclusion Criteria (melanoma):

* Histologically or cytologically documented findings consistent with advanced melanoma not amenable to curative surgery, radiation, or other therapy. Uveal melanoma is excluded.
* Patients who are not candidates for or have refused available therapies are also eligible.
* Received an anti-programmed death-1 (PD-1) / programmed death ligand-1 (PD-L1) inhibitor as monotherapy or in combination with anti-cytotoxic lymphocyte associated protein 4 (CTLA-4) inhibitor and have either primary or secondary checkpoint inhibitor resistance as per Society for Immunotherapy of Cancer (SITC) consensus definition, unless deemed intolerable by the investigator. Patients with BRAF V600E mutant melanoma should have received a BRAF inhibitor as monotherapy or in combination with other targeted agents (mitogen-activated protein kinase [MAPK] kinase [MEK] inhibitors), unless deemed intolerable by the investigator.
* Has disease other than the injected lesion that is measurable by RECIST 1.1.

Phase 1 and 2 Exclusion Criteria:

* History of primary immune deficiency.
* History of autoimmune disease and/or requiring immunosuppression (except hypothyroidism).
* History of History of Grade 3 or higher immune-related adverse events. Patient may be enrolled with Medical Monitor approval.
* History of solid organ transplant and taking immunosuppressive medications.
* Cardiovascular exclusions: Medical history of an arterial thrombotic event, stroke, or transient ischemic attack within the past 12 months; medical history of symptomatic congestive heart failure (New York Heart Association classes II-IV) or a cardiac arrhythmia that required treatment within the past 12 months; medical history of myocardial infarction or unstable angina within 6 months before Cycle 1 Day 1; QTcF prolongation to > 470 ms in women and > 450 ms in men based on a 12-lead electrocardiogram (ECG) in triplicate using the Fridericia formula: QTc = QT / RR1/3.

Recent medical concerns exclusions:

* Prior direct radiation therapy to the tumor lesion to be injected.
* Active use of systemic anticoagulants
* Evidence of active infection requiring intravenous (IV) antibiotics during screening requiring therapy within 7 days prior to Cycle 1 Day 1.
* Active uncontrolled bleeding, or a bleeding diathesis within 7 days prior to Cycle 1 Day 1.
* Serious or non-healing wound, fistula, skin ulcer, or non-healing bone fracture within 7 days prior to Cycle 1 Day 1.
* Known human immunodeficiency virus (HIV) infection, active hepatitis B infection, or hepatitis C infection.
* Virology evaluation should be conducted at screening to include serum HIV antibody, HBc antibody, HBsAg antigen, and HCV antibody. Patients with a positive antibody evaluation for HCV and/or HBc should undergo evaluation to measure HCV RNA or HBV DNA, respectively.
* Untreated central nervous system tumor, epidural tumor or metastasis, or brain metastasis. Patients with any primary Central Nervous System (CNS) malignancy including glioma and current, active, progressing CNS malignancy, including carcinomatosis meningitis are excluded.
* Patients with treated brain metastases are eligible if there is no evidence of progression for at least 4 weeks after CNS-directed treatment, as ascertained by clinical examination and brain imaging (magnetic resonance imaging [MRI] or computed tomography [CT] scan) during the screening period and off systemic steroids (for at least 2 weeks prior to first dose).
* Another primary malignancy that has not been treated with curative intent, except for non-metastatic cutaneous basal cell or squamous cell carcinoma, or non-muscle invasive bladder cancer.
* Serious illness considered by the Investigator as incompatible with participating in this clinical study.
* Any condition that, in the opinion of the Investigator, would interfere with evaluation of the investigational product or interpretation of the patient's safety or study results.
* Prior IL-12 therapy.
* Receipt of any vaccine within 30 days prior to the first dose of study treatment.
* Use of another anticancer therapy within 3 weeks prior to Cycle 1 Day 1 or 5 half-lives, whichever is shorter.
* Previously enrolled in this study.
* Actively enrolled in another clinical study unless it is an observational (noninterventional) clinical study or the follow-up component of an interventional study.
* Known severe hypersensitivity (Grade ≥ 3) to study treatment or any of the excipients of the products.
* Known psychiatric or substance use disorder that would interfere with the participant's ability to cooperate with the requirements of the study.
* Currently pregnant (confirmed with positive pregnancy test), breast-feeding or planning to become pregnant within 60 days following treatment. For women of childbearing potential (WOCBP), a negative serum beta-human chorionic gonadotropin (β-HCG) result must be available within a 72 hour window before the first treatment dose.
* Women of childbearing potential not willing to use a highly effective method of contraception.
* Unwilling or unable to follow protocol requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Estimated)
Dates: Start 2024-05-03 (Actual); Primary Completion 2027-05 (Estimated); Study Completion 2028-11 (Estimated)

PRIMARY OUTCOMES:
Number and nature of dose-limiting toxicities (DLTs), treatment-emergent adverse events (TEAEs) and serious adverse events (SAEs) in patients with advanced solid tumors. | From time of informed consent until 30 days after the last dose of investigational product (STX-001).
  The occurrence of DLTs, TEAEs, and SAEs will be used to determine the maximum tolerated dose and recommended Phase 2 dose of STX-001.
Occurrence of changes from baseline in patients' clinical safety laboratory values and vital signs to assess the safety and tolerability of STX-001. | From time of informed consent until 30 days after the last dose of investigational product (STX-001).
  Collection and analysis of changes in data from baseline of patients' vital signs (temperature, pulse, respiratory rate, blood pressure, oxygen saturation via pulse oximetry) as well as clinical safety laboratory values (chemistry, hematology, coagulation, complement (Bb & C3a), urinalysis, and lipids).

SECONDARY OUTCOMES:
Assessment of PK in patients dosed with STX-001 | From time of informed consent until 30 days after the last dose of investigational product (STX-001).
  Individual and mean plasma STX-001 concentrations versus time data will be collected, summarized, and plotted by dose level.
Assessment of Tumor infiltrating lymphocytes (TILs) | From time of informed consent until 30 days after the last dose of investigational product (STX-001).
  Assessment of STX-001 PK concentrations in mono therapy and safety and tolerability of STX-001 in combination with pembrolizumab in the tumor microenvironment (biopsy).
Number and nature of preliminary antitumor activity of STX-001. | From time of informed consent until 30 days after the last dose of investigational product (STX-001).
  Proportion of patients with objective response rate (ORR), complete response (CR), or partial response (PR) per RECIST 1.1.
Number and nature of preliminary antitumor activity of STX-001 in combination with pembrolizumab. | From time of informed consent until 30 days after the last dose of investigational product (STX-001).
  Proportion of patients with objective response rate (ORR), disease control rate (DCR), complete response (CR), partial response (PR) or stable disease (SD) per RECIST 1.1.
Number and nature of preliminary antitumor activity of STX-001. | From time of informed consent until 18 months after the last dose of investigational product (STX-001).
  Proportion of patients with progression-free survival (PFS), defined as the time from randomization to first evidence of radiographically detectable disease or death from any cause. Proportion of patients with duration of response (DOR) (CR or PR), per RECIST 1.1.
Number and nature of preliminary antitumor activity of STX-001 in combination with pembrolizumab. | From time of informed consent until 18 months after the last dose of investigational product (STX-001).
  Proportion of patients with progression-free survival (PFS), defined as the time from randomization to first evidence of radiographically detectable disease or death from any cause. Proportion of patients with overall survival (OS, duration of response (DOR) (CR or PR), per RECIST 1.1.
Occurrence of TEAEs, SAEs, and AESIs graded according to NCI CTCAE v5.0 | From time of informed consent until 30 days after the last dose of investigational product (STX-001).
  Assessment of the safety and tolerability of STX-001 in patients with advanced solid tumors.
Occurrence of changes from baseline in patients' clinical safety laboratory values and vital signs to assess the safety and tolerability of STX-001.in combination with pembrolizumab. | From time of informed consent until 30 days after the last dose of investigational product (STX-001).
  Collection and analysis of changes in data from baseline of patients' vital signs (temperature, pulse, respiratory rate, blood pressure, oxygen saturation via pulse oximetry) as well as clinical safety laboratory values (chemistry, hematology, coagulation, complement (Bb & C3a), urinalysis, and lipids).
Objective Response Rate (ORR) in patients with advanced solid tumors. | From time of informed consent until 30 days after the last dose of investigational product (STX-001).
  Objective Response Rate (ORR) is defined as the proportion of patients with confirmed response (CR) or confirmed partial response (PR).

CONTACTS AND LOCATIONS:
Overall Officials: Jason Luke, MD, Study Chair — Strand Therapeutics
Locations (7):
- United States (6):
  - HonorHealth Research and Innovation Institute, Scottsdale, Arizona
  - NextGen Oncology, Beverly Hills, California
  - Cleveland Clinic, Cleveland, Ohio
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
  - Huntsman Cancer Institute - University of Utah, Salt Lake City, Utah
- Melanoma Institute Australia, Wollstonecraft, Australia

IPD SHARING:
Plan to Share IPD: No